CLINICAL TRIAL: NCT03220919
Title: Efﬁcacy and Safety of Weight-Based Insulin Titration (WEB-IT) Regimen Compared With Glucose Level-based Regimen in Hospitalized Patients With Type 2 Diabetes: A Randomized Controlled Study
Brief Title: Efﬁcacy and Safety of Weight-Based Insulin Titration Regimen in Hospitalized Patients With Type 2 Diabetes
Acronym: WEB-IT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: weightbased
Record Dates: First submitted 2017-07-08; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Efficacy, Self; Adverse Effect
Keywords: Insulin; Type 2 diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-based (Experimental): Weight-based insulin insulin titration regimen
  Interventions: Other: Weight-based
- Glucose level-based (Placebo Comparator): Glucose level-based insulin titration regimen
  Interventions: Other: Glucose level-based

INTERVENTIONS:
Other: Weight-based — Glargine titration: 0.1U/kg per day when FBG is over 8.0 mmol/L. Aspart titration: total dose 0.1U/kg per day when next pre-meal BG is over 8.0 mmol/L, which is divided into three equal parts adding to three pre-meal boluses
  Arms: Weight-based
Other: Glucose level-based — Glargine titration: 4, 6, or 8 U when FBG is, respectively, within the following ranges: 8.0-8.9, 9.0-9.9, >10.0 mmol/L.
  Aspart titration: 1, 3, 5, 7 or 8 U when next pre-meal BG is, respectively, within the following ranges: 8.0-10.9, 11.0-13.9, 14.0-16.9, 17.0-19.9, > 20 mmol/L.
  Arms: Glucose level-based

SUMMARY:
The investigators propose to use a weight-based regimen consisting of basal-bolus insulin and preprandial rapid-acting insulin and to test its efficacy and safety in controlling blood glucose in hospitalized patients with type 2 diabetes.

DETAILED DESCRIPTION:
Patients with type 2 diabetes are randomly assigned by computer-generated block randomization to receive either weight-based or glucose level-based titration regimen. All antidiabetic drugs are discontinued on admission.

Starting dose:

Total daily insulin is 0.4U/kg. Half is given as glargine and the remainder as aspart which is divided into three equal parts used for three pre-meal boluses.

Titration:

1. Weight-based insulin titration regimen:

   Glargine titration: 0.1U/kg per day when fasting blood glucose (FBG) is over 8.0 mmol/L.

   Aspart titration: total dose 0.1U/kg per day when next pre-meal blood glucose (BG) is over 8.0 mmol/L, which is divided into three equal parts adding to three pre-meal boluses.
2. Glucose level- based titration regimen:

Glargine titration: 4, 6, or 8 U when FBG is, respectively, within the following ranges: 8.0-8.9, 9.0-9.9, >10.0 mmol/L.

Aspart titration: 1, 3, 5, 7 or 8 U when next pre-meal BG is, respectively, within the following ranges: 8.0-10.9, 11.0-13.9, 14.0-16.9, 17.0-19.9, > 20 mmol/L.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years with type 2 diabetes admitted to Endocrinology wards.

Exclusion Criteria:

* Patients with hepatic or renal dysfunction, cancer, or diabetic ketoacidosis;
* Patients who are pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Duration | at discharge, an average of 9 days
  Duration to achieve BG targets, including three pre-meal BG and bedtime BG
Doses | at discharge, an average of 9 days
  Doses of insulin glargine and insulin aspart when the BG targets are achieved

SECONDARY OUTCOMES:
Hypoglycemia | at discharge, an average of 9 days
  Incidence of hypoglycemia

OTHER OUTCOMES:
Adverse effects | at discharge, an average of 9 days
  Other adverse effects except hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Wangen Li, MD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang X, Zhang T, Xiang G, Wang W, Li Y, Du T, Zhao Y, Mosha SS, Li W. Comparison of weight-based insulin titration (WIT) and glucose-based insulin titration using basal-bolus algorithm in hospitalized patients with type 2 diabetes: a multicenter, randomized, clinical study. BMJ Open Diabetes Res Care. 2020 Sep;8(1):e001261. doi: 10.1136/bmjdrc-2020-001261. PMID 32933950